CLINICAL TRIAL: NCT07373990
Title: Short-course Tislelizumab Combined With Chemoradiotherapy for Locoregionally Advanced Nasopharyngeal Carcinoma: A Randomized, Controlled, Multicenter, Phase 3 Non-inferiority Clinical Trial
Brief Title: Short-course Tislelizumab Combined With Chemoradiotherapy for Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-462-FLK
Record Dates: First submitted 2025-12-29; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Nasopharyngeal Cancer
Keywords: tislelizumab; PD-1 antibody; short-course
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — tislelizumab; Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tislelizumab (3×200 mg q3w neoadjuvant + 3×400 mg q6w adjuvant) (Experimental): Patients will receive neoadjuvant gemcitabine (1000 mg/m2 d1, d8), cisplatin (80 mg/m2 d1) and tislelizumab (200 mg) every 3 weeks for 3 cycles, followed by defnitive intensitymodulated radiotherapy (IMRT) of 6996cGy in 33 fractions. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Subsequently, adjuvant therapy with tislelizumab (400 mg) every 6 weeks for 3 cycles.
  Interventions: Drug: tislelizumab; Drug: Gemcitabine + cisplatin (GP); Drug: Cisplatin (100mg/m2); Radiation: intensity-modulated radiotherapy
- tislelizumab (3×200 mg q3w neoadjuvant + 5×400 mg q6w adjuvant) (Active Comparator): Patients will receive neoadjuvant gemcitabine (1000 mg/m2 d1, d8), cisplatin (80 mg/m2 d1) and tislelizumab (200 mg) every 3 weeks for 3 cycles, followed by defnitive intensitymodulated radiotherapy (IMRT) of 6996cGy in 33 fractions. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Subsequently, adjuvant therapy with tislelizumab (400 mg) every 6 weeks for 5 cycles.
  Interventions: Drug: tislelizumab; Drug: Gemcitabine + cisplatin (GP); Drug: Cisplatin (100mg/m2); Radiation: intensity-modulated radiotherapy

INTERVENTIONS:
Drug: tislelizumab — Neoadjuvant tislelizumab 200 mg, every 3 weeks for 3 cycles; Adjuvant tislelizumab 400 mg, every 6 weeks for 3 cycles.
  Arms: tislelizumab (3×200 mg q3w neoadjuvant + 3×400 mg q6w adjuvant)
Drug: tislelizumab — Neoadjuvant tislelizumab 200 mg, every 3 weeks for 3 cycles; Adjuvant tislelizumab 400 mg, every 6 weeks for 5 cycles.
  Arms: tislelizumab (3×200 mg q3w neoadjuvant + 5×400 mg q6w adjuvant)
Drug: Gemcitabine + cisplatin (GP) — neoadjuvent gemcitabine (1000 mg/m2 d1, d8) and cisplatin (80 mg/m2 d1) every 3 weeks for 3 cycles
Drug: Cisplatin (100mg/m2) — Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
Radiation: intensity-modulated radiotherapy — Defnitive intensity-modulated radiotherapy (IMRT) of 6996cGy will be given in 33 fractions.

SUMMARY:
This trial aim to explore whether short-course tislelizumab (3 cycles of 200 mg q3w in the induction phase and 3 cycles of 400 mg q6w in the consolidation phase) yields non-inferior event-free survival compared to long-course tislelizumab (3 cycles of 200 mg q3w in the induction phase and 5 cycles of 400 mg q6w in the consolidation phase) in patients with locoregionally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤65 years
2. Patients with histologically confirmed non-keratinizing nasopharyngeal carcinoma according to WHO criteria.
3. Eastern Cooperative Oncology Group performance score of 0-1.
4. Tumor staged as T4N1 and T1-4N2-3 disease (AJCC 9th edition).
5. Adequate marrow function:

   white blood cell count > 4 × 10⁹/L hemoglobin >90g/L and platelet count >100×10⁹/L
6. Adequate hepatic and renal function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN), Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×ULN, Alkaline phosphatase ≤ 2.5 ×ULN, clearance rate ≥ 60 ml/min 7. Other laboratory and clinical criteria Normal: thyroid function, serum amylase and lipase, pituitary hormone levels, inflammatory markers, cardiac enzyme tests and electrocardiogram (ECG); For patients aged >50 years with a history of smoking, normal pulmonary function test (PFT) results are required; For patients with abnormal ECG findings or a prior history of cardiovascular disease (not meeting any exclusion criteria listed in Item 8), additional assessments including myocardial function evaluation and cardiac ultrasound (echocardiography) must be performed, with results within normal limits.

8. Patients must be informed of the investigational nature of this study and give written informed consent, and be willing and able to comply with the study schedule, including follow-up visits, treatment procedures, laboratory testing, and other protocol-related requirements.

9. Women of childbearing potential (WOCBP) must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen (HBsAg) with hepatitis B virus DNA >1×10 copies/mL, positive for anti-hepatitis C virus (HCV) antibody, positive for anti-hepatitis C virus (HCV) antibody
2. Positive for anti-HIV antibody or diagnosed with acquired immunodeficiency syndrome (AIDS).
3. Active pulmonary tuberculosis: Patients with a history of active tuberculosis within the past year should be excluded regardless of treatment status. Patients with a history of active pulmonary tuberculosis more than one year prior should also be excluded, unless they received con dirmed and regular anti-tuberculosis treatment.
4. Active, known, or suspected autoimmune diseases, including but not limited to uveitis, colitis, hepatitis, hypophysitis, nephritis, vasculitis, systemic lupus erythematosus, hyperthyroidism, hypothyroidism, and asthma requiring bronchodilators. Type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) are allowed.
5. History of interstitial lung disease or pneumonia requiring oral or intravenous corticosteroids within the past year; use of vancomycin within the past month.
6. Ongoing chronic systemic corticosteroid therapy (equivalent to or greater than prednisone >10mg per day) or any other immunosuppressive therapy. Patients received inhale or topical corticosteroid are allowed.
7. Uncontrolled cardiac conditions, such as: Heart failure with New York Heart Association (NYHA) classi dication ≥ Class II; or Unstable angina; or History of myocardial infarction within the past year; or Supraventricular or ventricular arrhythmias requiring treatment or intervention
8. Pregnant or breastfeeding women (pregnancy testing should be considered for women of childbearing potential with active sexual life)
9. History or presence of other malignancies, except for adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary thyroid carcinoma.
10. Known hypersensitivity to macromolecule protein products.
11. Active infections requiring systemic treatment within 1 week prior to enrollment.
12. Administration of live vaccines within 30 days prior to the first dose of tile.
13. History of organ transplantation or hematopoietic stem cell transplantation.
14. Any other condition assessed by the investigator as potentially compromising patient safety or compliance, such as severe illnesses requiring urgent treatment (including psychiatric disorders), significantly abnormal laboratory values, or other psychological, familial, or social risk factors.
15. Patients who have previously received immune checkpoint (CTLA-4, PD-1, PD-L1, etc.) inhibitor therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3 years
  From date of randomization until the date of first documented locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  From date of randomization until the date of death from any cause, whichever came first
Distant metastasis-free survival (DMFS) | 3 years
  From date of randomization until the date of first documented distant metastasis, whichever occurred first
Locoregional recurrence-free survival (LRRFS) | 3 years
  From date of randomization until the date of first documented locoregional recurrence, whichever occurred first
Adverse events (AEs) | within 5 years
  Graded according to CTCAE V5.0
Quality of life (QoL) | week 0, 9, 16, 28, 40 and 1 year, 2 years, 3 years, 4 years, and 5 years after randomization
  The EORTC QoL questionnaire-C30 (EORTC QLQ-C30）version 3.0 will be used.The change of QoL from randomization to 9 weeks (at the end of neoadjuvant treatment), 16 weeks (at the end of radiotherapy), 28 weeks (at the 3nd cycle of adjuvant tislelizumab treatment), 40 (at the 5nd cycle of adjuvant tislelizumab treatment, if available), 1 year, 2 years, 3 years, 4 years, and 5 years after randomization. This questionnaire comprises 30 questions, 24 aggregated into nine multi-question scales: five functioning scales (e.g., physical), three symptom scales (e.g., fatigue), and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual of EORTC QLQ-C30.
cost-effectiveness analysis | 3 years
  Cost-effectiveness will be evaluated as the incremental cost per clinical outcome achieved (e.g., cost per quality-adjusted life year gained or cost per event avoided) when comparing the intervention and control groups.

IPD SHARING:
Plan to Share IPD: No